CLINICAL TRIAL: NCT07364656
Title: Analysis of the Presence and Cardiac Functional Effects of Anti-NaV1.5 Autoantibodies in Patients With Metastatic Tumors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Policlinico S. Donato (Other)
Collaborators: IRCCS San Raffaele (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NAV-CARD
Record Dates: First submitted 2026-01-09; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-10

CONDITIONS: Brugada Syndrome (BrS); Breast Cancer Females; Colon Cancer; ECG Abnormalities; Autoantibodies Screening
MeSH Terms: conditions — Brugada Syndrome; Colonic Neoplasms | interventions — Electrocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- breast cancer (Other)
  Interventions: Diagnostic Test: ECG
- metastatic brest cancer (Other)
  Interventions: Diagnostic Test: ECG
- colon cancer (Other)
  Interventions: Diagnostic Test: ECG
- metastatic colon cancer (Other)
  Interventions: Diagnostic Test: ECG

INTERVENTIONS:
Diagnostic Test: ECG — These patients require an ECG to exclude the onset of arrhythmias.

SUMMARY:
The overall aim of this study is to identify and characterize anti-NaV1.5 autoantibodies in patients with metastatic breast and colorectal cancer. These tumors are characterized by the presence of a specific target structure (called nNaV1.5) against which antibodies are produced. These antibodies may cross-react with a similar structure (called NaV1.5) that is found in the heart. This could affect channel function and increase the risk of arrhythmias.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients with a confirmed diagnosis of breast or colorectal cancer, either metastatic or non-metastatic
* Patients already receiving first-line therapy with a confirmed diagnosis of breast or colorectal cancer, either metastatic or non-metastatic
* Signed informed consent

Exclusion Criteria:

* Clinically significant cardiovascular diseases (atrial fibrillation, congestive heart failure, cardiomyopathies, or inherited arrhythmic syndromes)
* Known autoimmune diseases or immunodeficiencies
* Use of high-dose immunosuppressive drugs or other experimental treatments that could interfere with the assessment of study endpoints

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Presence of circulating autoantibodies against SCN5A in plasma of enrolled patients, assessed at baseline (enrollment) and at 6- and 12-month follow-up visits. | Baseline (at enrollment), 6 months, and 12 months.
  The primary outcome of this study is the detection of circulating autoantibodies against the cardiac sodium channel SCN5A in the plasma of enrolled patients. Plasma samples will be collected at baseline, corresponding to study enrollment, and during follow-up visits at 6 and 12 months. The presence or absence of anti-SCN5A autoantibodies will be assessed to evaluate their prevalence and persistence over time and to explore their potential association with disease mechanisms and progression.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico San donato, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data including demographic characteristics, clinical variables relevant to the study, and laboratory results related to the presence or absence of anti-SCN5A autoantibodies at baseline, 6-month, and 12-month follow-up assessments.